CLINICAL TRIAL: NCT00185510
Title: Double-Blind, Placebo Controlled, Randomized, Multicenter, Parallel-Group Study to Compare the Efficacy and Safety of Advantan Cream Twice Weekly With Advabase Cream During a Maintenance Phase of 16 Weeks After Successful Treatment of Atopic Dermatitis With Advantan Cream
Brief Title: Efficacy and Safety Study of Advantan for Maintenance Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91424; 2004-002673-22 (EudraCT Number); 309189 (Other: Company internal)
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2014-02

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — methylprednisolone aceponate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Methylprednisolone Aceponate (Advantan, BAY86-4862)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone Aceponate (Advantan, BAY86-4862) — In maintenance phase, Methylprednisolone Aceponate cream is applied topically twice a week.
  Arms: Arm 1
Drug: Placebo — 2 days a week Vehicle (Advabase)
  Arms: Arm 2

SUMMARY:
Purpose of the study:

One bothering feature of atopic dermatitis is its relapsing nature. Hence, it is worthwhile to test modes how to efficiently prevent relapses or at least increase the time until the disease recurs. In order to give recommendations to other patients, this study is to scientifically describe efficacy and safety of a given regimen, namely a maintenance therapy with two days a week Advantan.

DETAILED DESCRIPTION:
The study has initially been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Intendis GmbH, a Bayer HealthCare company, is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute 'Severe' or 'Very Severe' flare of atopic dermatitis; no minimum affected body surface
* History of moderate to severe form of atopic dermatitis for at least two years

Exclusion Criteria:

* Pregnancy, breast feeding
* Known immune, hepatic, or renal insufficiency
* Acute herpes simplex or mollusca contagiosa infection
* Acute and severe impetigo contagiosa. A slight superinfection of eczema is no exclusion criterion
* Severe other viral, bacterial, or fungal skin infection (chicken pox, prominent tinea corporis)
* Acute infestations (e.g. head lice, scabies)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Time to relapse in the maintenance phase (MP) | Week 16

SECONDARY OUTCOMES:
Patients' number of relapses in the maintenance phase | Week 16
Treatment success as assessed by Investigator Global Assessment (IGA) score | Week 16
Percentage change during Acute Phase (AP) and MP assessed by Modified Eczema Area and Severity Index (mEASI) | Week 16
Index lesion monitoring | Week 16
Change of disease during AP and MP as assessed by Patient Global Assessment | Week 16
Visual assessment of signs of atrophy | Week 16
Ultrasound for measurement of skin thickness in selected sites | Up to week 16
Dermatology Life Quality Index (CDLQI, DLQI) | Week 16
Adverse Event Collection | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer